CLINICAL TRIAL: NCT00914017
Title: Statins and Breast Cancer Biomarkers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Collaborators: Breast Cancer Research Foundation (Other); Cancer and Leukemia Group B (Network)
Responsible Party: Marie Wood, MD, Vermont Cancer Center at University of Vermont and Fletcher Allen Health Care
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V0407; CHRMS#: 05-059
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2010-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast Cancer Prevention; Mammographic Density; Breast Density; Breast Cancer Biomarkers
MeSH Terms: conditions — Breast Neoplasms | interventions — Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Experimental): 40 mg of Lipitor (atorvastatin) daily for 1 year
  Interventions: Drug: Atorvastatin
- Sugar Pill (Placebo Comparator): Sugar pill daily for 1 year
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin, 40 mg daily for 1 year
  Other Names: Lipitor; statin
  Arms: Atorvastatin
Drug: Placebo — sugar pill daily for 1 year
  Arms: Sugar Pill

SUMMARY:
There is laboratory evidence that cholesterol lowering medications (statins) inhibit the growth of breast cancer cells. Clinical studies are controversial but some show that women taking statins are less likely to get breast cancer. This ongoing randomized trial compares one-year of atorvastatin (Lipitor™) or placebo for lowering mammography-defined breast density and other surrogate markers associated with breast cancer risk.

DETAILED DESCRIPTION:
This project was designed to evaluate the effect of a specific statin (atorvastatin) on several breast cancer biomarkers. One hundred women will be treated for one year with either 40 mg of atorvastatin or placebo. The primary aim of this project is to determine the effect of atorvastatin on breast density, a known risk factor for breast cancer. In addition, the affect of atorvastatin on serum biomarkers (IGF1) and tissue biomarkers (atypia and Ki67) associated with risk is being evaluated.

Because of their tolerability and safety, statins have a great potential as a breast cancer preventative agent. Should this pilot study show a significant decrease in breast density and/or change in serum and tissue biomarkers in statin treated patients these data would then be used to support a large randomized trial.

This is a multi-center, prospective, randomized placebo controlled clinical trial. Target enrollment is 100 women, with 50 receiving atorvastatin and 50 receiving a similar appearing placebo tablet. Eligible women must be at least 35 years old with regular menstrual cycles and a Gail Model risk of greater than 1.66% over 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Women willing and able to give written informed consent
* Pre-menopausal women with regular menstrual cycles (4 cycles in the past 6 months)
* At least 35 years of age
* Women at increased risk of developing breast cancer, defined as at least one of the following four criteria:

  * Having had a biopsy demonstrating atypical hyperplasia or lobular neoplasia/LCIS
  * A germline mutation in BRCA1/2 in themselves or their family.
  * A Gail Model Risk of > 1.67% over 5 years
  * A strong family history of breast and/or ovarian cancer which is defined as at least one of the following:

    * One first-degree relative with breast cancer before the age of 50 years
    * One first degree relative with bilateral breast cancer
    * Two or more first-degree relatives with breast cancer
    * One first degree relative and two or more second or third degree relatives with breast cancer
    * One first-degree relative with breast cancer and one or more relatives with ovarian cancer
    * Two second or third degree relatives with either breast cancer and one or more with ovarian cancer
    * One second or third degree relative with breast cancer and two or more with ovarian cancer
    * Three or more second or third degree relatives with breast cancer
  * A prior history of breast cancer, including DCIS and stage 0-IIIb, and are at least one year off of all therapy (including radiation, biologic, hormonal and/or chemotherapy)

Exclusion Criteria:

* Women with a prior history of stage IV breast cancer or ovarian cancer
* Women already taking statins. Women previously on statins may participate if they have not taken any statins in the six months prior to study entry
* Women concurrently participating in another breast cancer chemoprevention trial
* Women taking hormone replacement therapy (estrogen and progesterone; topical estrogen will be allowed)
* Women taking tamoxifen, raloxifene, or an aromatase inhibitor
* Women taking drugs that increase risk of statin induced myopathy or rhabdomyolysis (i.e., Niacin, protease inhibitors, verapamil, gemfibrozil, cyclosporine, clofibrate/fenofibrate or any CYP3A4 inhibitor)
* Women with underlying liver disease or abnormal liver studies including:

  * alkaline phosphatase, ALT, AST and Bilirubin (greater than 1.5 times normal)
* Women who have had hypersensitivity to atorvastatin or any component of the formulation
* Women who are pregnant, planning pregnancy within the next year, or breastfeeding

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-01; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate change in percent mammographic density after one year of statin administration in pre-menopausal women at high risk for breast cancer. | 1 year

SECONDARY OUTCOMES:
To evaluate changes in IGF1 levels after 12 months of statin administration in pre-menopausal women at high-risk for breast cancer. | 1 year
To correlate changes in breast density with changes in molecular markers. | 1 year
To explore changes in breast duct cell cytology in a subset of patients after 12 months of statin administration in a subset of the trial population. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marie E Wood, MD, Principal Investigator — University of Vermont
Locations (7):
- United States (7):
  - University of California, San Francisco, San Francisco, California
  - Delaware Christiana Care CCOP, Helen F. Graham Cancer Center, Newark, Delaware
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Duke University, Durham, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Vermont Cancer Center, Burlington, Vermont

REFERENCES:
- See also: High Risk Breast Program of Vermont, Research Studies — http://hrbp.vermontcancer.org/?page_id=4